CLINICAL TRIAL: NCT06372392
Title: Randomized Controlled Study of the Usage of Universal Fixed Meal Bolus Coefficients for the Control of Postprandial Hyperglycemia in the Users of Medtronic Minimed 780G Pumps
Brief Title: Universal Fixed Meal Boluses Usage in Patients With Medtronic Minimed 780G Pumps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Collaborators: Estonia Research Council (Unknown)
Responsible Party: Principal Investigator, Aleksandr Peet, Pediatric endocrinologist (PI), Tartu University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2024-04-10; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Type1diabetes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Universal coefficient (Experimental): With fixed meal bolus coefficients (TDD/300 breakfast and TDD/400 other meals)
  Interventions: Device: Universal meal coefficient utilization
- Individualized coefficient (Active Comparator): With meal bolus coefficient individualized according to physician judgment's
  Interventions: Device: Universal meal coefficient utilization

INTERVENTIONS:
Device: Universal meal coefficient utilization — Usage of universal fixed meal bolus coefficients for the control of postprandial hyperglycemia compared to individualized coefficients n the users of Medtronic Minimed 780G pumps

SUMMARY:
Cross-over study of 20 pediatric patients (age 7-19) randomized to the group receiving universal fixed meal boluses coefficients (300/TDD for breakfast and 400/TDD other meal) or to the group with individualized coefficients for the period of 14 days with consecutive analysis of the results from Carelink Raport.

ELIGIBILITY:
Inclusion Criteria:

* age 7-19
* type 1 diabetes diagnosed at least 1 year ago
* insulin in the dose 0,5-1,0 units/day/kg
* MiniMed 780G pump usage at least 1 month.

Exclusion Criteria:

* Active coeliac disease
* Chronic disease possible to influence diabetes treatment
* Acute disease at the moment of recruitment

Ages: 7 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Time in range (TIR) | 4 weeks
  Comparision of TIR between groups

SECONDARY OUTCOMES:
TBR | 4 weeks
  Comparision of TBR between groups
TAR | 4 weeks
  Comparision of TAR between groups
auto-corrections % | 4 weeks
  auto-corrections % between groups
coefficient of variability | 4 weeks
  coefficient of variability between groups

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Peet, Principal Investigator — Tartu University Hospital
Locations (1):
- TartuUH, Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No